CLINICAL TRIAL: NCT06878157
Title: Ontological Coaching Among Novice Nurses (OCN): a Mixed Methods Study
Brief Title: Ontological Coaching Among Nurses (OCN)
Acronym: OCN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Shefaly Shorey, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NHG DSRB 2022/00676
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Ontological Coaching; Psychological Wellbeing

STUDY DESIGN:
Intervention Model Description: Two-group parallel-armed randomized controlled trial with an intervention group undergoing ontological coaching and control group with no ontological coaching.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coaching (Experimental): In the form of small groups (3-6 participants), the nurses will receive a knowledge based session (maximum 1 hour long) to share about ontological coaching. After the group session, each nurse will receive 4 individual sessions (30-60 minutes) on monthly basis.
  Interventions: Behavioral: ontological coaching
- Conotrol (No Intervention): Participants do not undergo any ontological coaching.

INTERVENTIONS:
Behavioral: ontological coaching — Group session: This session will provide an overview of coaching and the following topics will be covered: 1) Experience coaching in teams, 2) The Ideal Life, 3) The Coaching Distinction, 4) Introduction to Body, Emotions, Language (BEL), 5) Deeper understanding of BEL, 6) Applying BEL to clinical scenarios, 7) The coaching perspective in Nursing, 8) Re-visit the Ideal Life, 9) Explore mental/emotional/physical challenges in practicing nursing, 10) Time and stress management, work-life balance; Individual Session: This individualized session will cover the discussions on the topic brought up by novice nurses. The aim of this session is to: 1) Help novice nurses design the steps in their journey towards what they care about, 2) Explore the nurses' world by asking encouraging and evoking questions, 3) Collaborate with nurses in a stimulating and imaginative manner that help them to optimize their potential, 4) Co-create with nurses the professional and personal identity they strive for
  Arms: Coaching

SUMMARY:
This study aims to develop and evaluate ontological coaching among novice nurses in Singapore. The specific aims of this project are: (1) to develop theory based Ontological Coaching among Nurses (OCN) intervention for novice nurses; (2) examine its effectiveness on nurses' psychological wellbeing (primary outcome), help-seeking behavior (social support), goal setting, resilience, intention to leave and job satisfaction (Secondary outcomes); and (3) examine the perceptions of nurses in receiving this intervention.

The specific research questions we plan to answer in this project are:

* How the OCN will influence psychological wellbeing of the new nurses?
* How the OCN will enhance the new nurses social support and goal setting for their reality and future?
* How the OCN will influence new nurses' resilience, intention to leave and job satisfaction?
* What are the changes in psychological well-being, social support, goal setting, resilience, intention to leave and job satisfaction after receiving OCN over time (pre-test and post-test)?
* Are there any strengths, weaknesses and area of improvements (overall experience) for the use of OCN among new nurses?

ELIGIBILITY:
Inclusion Criteria:

Nurses:

* 21 years old and above
* are able to read and speak English,
* have 0-10 years of working experience after the registration with Singapore Nursing Board (SNB)
* currently working at the study venues with the valid registered nurse license with the SNB
* who are willing to be audio-recorded if invited for an interview

Facilitators:

- who hold an Ontological Coaching certification and a minimum of 50 hours of Coaching experience

Exclusion Criteria:

Nurses:

* have physical or mental disorders which would interfere with their ability to participate in the study
* have refused to participate in this study

Facilitators:

- who does not hold an Ontological Coaching certification or who do not have a minimum of 50 hours of Coaching experience

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
Effectiveness on nurses' psychological wellbeing | baseline, 2-3 months (intervention), 4-6 months (post intervention)
  Ryff Scales of Psychological Well-Being: a 42-item instrument Psychological Wellbeing (PWB) Scale measures six aspects of wellbeing and happiness: autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance. Respondents rate how strongly they agree or disagree with 42 statements using a 7-point scale (1 = strongly agree; 7 = strongly disagree).

SECONDARY OUTCOMES:
Stress | baseline, 2-3 months (intervention), 4-6 months (post intervention)
  Nursing Stress Scale: a 34-item instrument that describe situations that have been identified as causing stress for nurses in the performance of their duties. Respondents how strongly they agree or disagree with 34 statements using a 4-point scale (1 = never; 4 = very frequently).
Help-seeking behavior (social support) | baseline, 2-3 months (intervention), 4-6 months (post intervention)
  Sarason's social support questionnaire - short form (SSQSR): a 6-item instrument to evaluate the availability and satisfaction associated with an individual's social support systems. Respondents indicate the number of people available to provide support in 6 areas and then rate the overall level of satisfaction with the support given in each of the areas using a 6-point scale (1 = very dissatisfied; 6 = very satisfied).
Goal Setting | baseline, 2-3 months (intervention), 4-6 months (post intervention)
  Goal Setting Questionnaire (GSQ): an 18-item instrument to evaluate individuals' competencies in three areas: setting meaningful goals, focusing on personal improvement, and incorporating prior experiences, interests, skills, and feedback from family, peers, or a trusted individual. Respondents rate how strongly they agree or disagree with 18 statements using a 5-point scale (1 = not very like me; 5 = very like me)
Intention to Leave | baseline, 2-3 months (intervention), 4-6 months (post intervention)
  Roodt's turnover scale (TIS-6): a 6-item instrument to measure turnover intention. Respondents rate how strongly they agree or disagree with 6 statements using a 5-point scale (1 = never; 5 = always)
Job Satisfaction | baseline, 2-3 months (intervention), 4-6 months (post intervention)
  Bowling Green State University's The Job Satisfaction Scale: measures employee attitudes such as job satisfaction. Respondents indicate their satisfaction in 5 areas (Y = Yes; N = No; ? = Cannot Decide).

CONTACTS AND LOCATIONS:
Overall Officials: Shefaly Shorey, PhD, Principal Investigator — National University of Singapore
Locations (4):
- Singapore (4):
  - Alexandra Hospital, Singapore
  - National University Hospital, Singapore
  - National University Polyclinics, Singapore
  - Ng Teng Fong General Hospital, Singapore